CLINICAL TRIAL: NCT00019019
Title: A PHASE I STUDY OF THE COMBINATION OF CAI AND PACLITAXEL IN ADULT PATIENTS WITH REFRACTORY CANCERS OR LYMPHOMA
Brief Title: Carboxyamidotriazole and Paclitaxel in Treating Patients With Advanced Solid Tumors or Refractory Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 950015; 95-C-0015; NCI-CPB-334; NCI-T94-0006N; CDR0000063881; NCT00001423 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors; Breast Cancer; Kidney Cancer; Lung Cancer; Lymphoma; Melanoma (Skin); Ovarian Cancer; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; recurrent adult brain tumor; small intestine lymphoma; adult brain stem glioma; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult glioblastoma; stage III melanoma; stage IV melanoma; recurrent melanoma; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IIIC breast cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult central nervous system germ cell tumor; primary central nervous system non-Hodgkin lymphoma; adult pilocytic astrocytoma; adult subependymoma; adult ependymoblastoma; adult pineocytoma; adult pineoblastoma; adult meningeal hemangiopericytoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; adult choroid plexus tumor; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult grade III meningioma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Breast Neoplasms; Kidney Neoplasms; Lung Neoplasms; Lymphoma; Melanoma; Ovarian Neoplasms; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Lymphoma, T-Cell, Cutaneous; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Brain Neoplasms; Craniopharyngioma; Medulloblastoma; Meningioma; Glioblastoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Pinealoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Choroid Plexus Neoplasms; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Gliosarcoma | interventions — carboxyamido-triazole; Paclitaxel

INTERVENTIONS:
Drug: carboxyamidotriazole
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of carboxyamidotriazole and paclitaxel in treating patients with advanced solid tumors or refractory lymphomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of paclitaxel when combined with carboxyamidotriazole in patients with advanced solid tumors or refractory lymphomas.
* Determine the pharmacokinetics and toxicities of this regimen in these patients.
* Identify diseases for which this combination appears active.

OUTLINE: This is a dose escalation study.

Patients receive oral carboxyamidotriazole (CAI) daily with paclitaxel IV over 3 hours on day 8 and every 3 weeks thereafter. Course 1 is 28 days and all other subsequent courses are 21 days. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response receive 2 additional courses of treatment.

Sequential dose escalation of CAI is followed by sequential dose escalation of paclitaxel. Dose escalation in cohorts of 3 to 6 patients each continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically diagnosed solid tumor (i.e., breast and ovarian epithelial carcinomas) or lymphoma

  * Slides reviewed at the NCI Laboratory of Pathology
* Failure on therapy of proven efficacy for the disease

  * Prior therapy not required for the following metastatic diseases:

    * Melanoma
    * Non-small cell lung cancer
    * Renal cell carcinoma
* No brain metastases

  * Primary brain tumors (such as glioblastoma multiforme) with stable neurologic deficits allowed
* Measurable or evaluable disease required

  * Demonstrated by physical exam or on radiograph within 2 weeks prior to initiation of treatment OR
  * Elevated PSA associated with prostate cancer

    * Other marker-only disease ineligible

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hematocrit at least 27%

Hepatic:

* Liver function tests no greater than 2 times upper limit of normal
* Bilirubin normal
* PT or PTT no greater than 1.25 times upper limit of normal
* Clotting parameters normal
* No concurrent anticoagulants other than 1 mg of warfarin per day for prophylaxis

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 45 mL/min
* No kidney obstruction

Cardiovascular:

* No cardiac conduction defect requiring antiarrhythmics
* No evidence of myocardial infarction or other myocardial damage within past 6 months

Other:

* HIV negative
* No concurrent infection
* No guaiac-positive stool test
* No neuropathy greater than grade I (unless associated with fixed-deficit primary brain tumors)
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

* Recovery from prior therapy required

Biologic therapy:

* At least 4 weeks since prior biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks since mitomycin, nitrosoureas, or carboplatin)
* No progression on carboxyamidotriazole or paclitaxel
* At least 6 months between treatment and relapse

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy
* No concurrent corticosteroids except as physiologic replacement

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 1 week since prior therapeutic antibiotics
* Concurrent prophylactic antibiotics allowed except imidazole antifungals (e.g., ketoconazole, fluconazole)
* No concurrent calcium channel blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 1994-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kwitkowski, MS, RN, CS, CRNP, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Medical Oncology Clinical Research Unit, Bethesda, Maryland

REFERENCES:
- [Result] Kohn EC, Reed E, Sarosy GA, Minasian L, Bauer KS, Bostick-Bruton F, Kulpa V, Fuse E, Tompkins A, Noone M, Goldspiel B, Pluda J, Figg WD, Liotta LA. A phase I trial of carboxyamido-triazole and paclitaxel for relapsed solid tumors: potential efficacy of the combination and demonstration of pharmacokinetic interaction. Clin Cancer Res. 2001 Jun;7(6):1600-9. PMID 11410496